CLINICAL TRIAL: NCT02381782
Title: Validation of uHear™ as a Screening Tool to Detect Hearing Impairment in Elderly Cancer Patients Within a Comprehensive Geriatric Assessment
Acronym: UHEAR
Status: Completed | Type: Observational
Sponsor: General Hospital Groeninge (Other)
Responsible Party: Principal Investigator, Dr. Philip Debruyne, Medical Oncologist, General Hospital Groeninge
Other Study IDs: AZGS2014125
Record Dates: First submitted 2015-03-05; First posted 2015-03-06 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Hearing Loss; Cancer
MeSH Terms: conditions — Hearing Loss; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Over the last few years, there has been a considerable interest in the development of screening tools to assess the capability of elderly cancer patients to tolerate anti-cancer treatment. Therefore, the NCCN Guidelines in Senior Adult Oncology recommend an assessment of co-morbid conditions that are likely to interfere with cancer treatment and tolerability. As presbyacusis is common in an older population, elderly cancer patients are at high risk for social isolation and a reduced quality of life. Therefore, in this project the investigators aim to validatie uHear™ as a quick and reliable screening tool to screen for presbyacusisf in routine clinical oncology practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients should have reached the age of 70 or more at enrolment
* Histologically confirmed diagnosis of solid cancer or hematologic malignancy. All stages of cancer are eligible
* Patients should be fluent in Dutch or French
* Patients must receive their primary oncology care in the participating hospital
* Patients should be cognitively capable of performing the audiology assessment
* Patients should have signed informed consent

Exclusion Criteria:

* Patients who do not match the above inclusion criteria
* Patients who are visiting the oncology clinic for a second opinion and do not wish to be treated in this clinic
* Patients presenting with clinically diagnosed Ménière's disease, retrocochlear hearing loss, autoimmune inner ear disease, fluctuating hearing loss or a history of sudden sensory neural hearing loss
* Patients who already have a hearing aid or a previously diagnosed hearing loss

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All consenting patients, aged ≥ 70, who are referred for anti-cancer treatment in the General Hospital Groeninge and who are in need of a CGA.
Sampling Method: Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2014-12; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Validation of uHear™ as a screening tool to detect hearing loss in elderly cancer patients | Baseline

SECONDARY OUTCOMES:
To determine the prevalence of presbyacusis in an elderly cancer population | Baseline
To compare objective and subjective hearing screening measures | Baseline
To measure hearing impairment in G8 positive patients compared with G8 negative patients | Baseline
To compare uHear™ with the Whispered Voice Test | Baseline
To evaluate the use of uHear™ as a measure to determine eligibility for cisplatin treatment in elderly cancer patients | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Philip R Debruyne, MD, PhD, Principal Investigator — Cancer Center, General Hospital Groeninge
Locations (1):
- General Hospital Groeninge, Kortrijk, Belgium

REFERENCES:
- [Result] Lycke M, Boterberg T, Martens E, Ketelaars L, Pottel H, Lambrecht A, Van Eygen K, De Coster L, Dhooge I, Wildiers H, Debruyne PR. Implementation of uHear--an iOS-based application to screen for hearing loss--in older patients with cancer undergoing a comprehensive geriatric assessment. J Geriatr Oncol. 2016 Mar;7(2):126-33. doi: 10.1016/j.jgo.2016.01.008. Epub 2016 Feb 26. PMID 26924571